CLINICAL TRIAL: NCT02793336
Title: Early Life Cohort in Papua Indonesia (ELIPI Study)
Acronym: ELIPI
Status: Completed | Type: Observational
Sponsor: Menzies School of Health Research (Other)
Collaborators: Timika Research Facility Kompleks RSMM, Timika-Papua, Indonesia (Unknown)
Responsible Party: Sponsor
Other Study IDs: ELIPI
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- infant cohort: The study is designed as a continuation of a cohort of infants from 12 to 48 months of age. This follows on from two previous cohorts: "STOP MIP", which is a cohort of pregnant women followed up until delivery and the "Baby-Cohort study", which enrols babies from mothers in the "STOP MIP" trial and follows them until their first year of live. When participants of the "Baby-cohort Study" reach study end, they are offered to participate in this study.

SUMMARY:
Malaria remains an important cause of illness in young infants. Our clinical and epidemiological studies in Papua (Indonesia) have shown the magnitude of malaria morbidity in infants in the first 5 years of life, including recurrent episodes of malaria, anaemia, malnutrition and coinfection. Together these contribute significantly morbidity in early life, and almost certainly to the very high infant mortality rates in this region. However the body of knowledge around infant malaria outside of Africa, where both species P. vivax and P. falciparum are prevalent is considerable smaller. The impact of recurrent vivax malaria and severe anaemia on neurodevelopment and growth in young children is unknown in Papua.

This study therefore aims to provide longitudinal data on the incidence of symptomatic and asymptomatic malaria (P. falciparum and P. vivax) and the associated risk of anaemia. It also provides an opportunity to assess incidence risk of non-malaria febrile illnesses and bacterial co-infections and the long term outcomes in terms of neurodevelopment and growth in a vulnerable age group. The study is a continuation from two already established cohort studies: "STOP MIP", which enrolled pregnant women and followed them until delivery and a "baby-cohort", which enrolled babies from mothers included in the cohort and followed them through their first year of life. Continuous follow up of those babies until they are 4 years old will increase our understanding of long term impact especially of vivax malaria. The cohort will be linked to a randomized controlled trial (RCT) and will offer cohort patients to be enrolled into the RCT when they are diagnosed with malaria (symptomatic), allowing to estimate treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patient enrolled in the Baby-Cohort study

Exclusion Criteria:

* Patients not enrolled in the Baby-Cohort study

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study is designed as a continuation of a cohort of infants from 12 to 48 months of age. This follows on from two previous cohorts: "STOP MIP", which is a cohort of pregnant women followed up until delivery and the "Baby-Cohort study", which enrols babies from mothers in the "STOP MIP" trial and follows them until their first year of live. When participants of the "Baby-cohort Study" reach study end, they are offered to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
P. vivax parasitaemia (PCR or microscopy) | 1 year
  The incidence rate of any P. vivax parasitaemia (PCR or microscopy) over 1 year in all infants

SECONDARY OUTCOMES:
symptomatic P. vivax | 1 year
  The incidence rate of symptomatic P. vivax over 1 year in all participants
severe anaemia (Hb<7g/dl) and/or blood transfusion | 4 years
  The incidence risk of severe anaemia (Hb<7g/dl) and/or the risk for blood transfusion
serious illnesses including hospitalization | 4 years
  The incidence risk and rate of serious illnesses including hospitalization
non-malarial febrile episodes and bacterial co-infections | 4 years
  The incidence risk and rate of non-malarial febrile episodes and bacterial co-infections
mortality | 4 years
  The incidence risk of mortality
growth retardation and neurodevelopment delay | 4 years
  The incidence risk of growth retardation and neurodevelopment delay
G6PD activity | 1 year
  The distribution of G6PD activity within the study population
Fluorescence spot test results (FST) | 1 year
  The change in FST result performed during the baby cohort study compared to the FST result performed at 12 months age

CONTACTS AND LOCATIONS:
Locations (1):
- Timika Research Facility, Timika, Timika-Papua, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided